CLINICAL TRIAL: NCT06745089
Title: Treatment Effect of Intense Pulsed Light and Thermal Pulsation Therapy on Meibomian Gland Dysfunction-associated Dry Eye Disease: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Nobel Eye Institute (Unknown); National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Wen-Chuan Kuo, Professor and Director, Institute of Biophotonics, National Yang Ming Chiao Tung University, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB number: YM111073F
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye Disease (DED); Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IPL arm (Experimental)
  Interventions: Device: Intense pulsed light
- TPT arm (Experimental)
  Interventions: Device: thermal pulsation therapy
- Control arm (Active Comparator)
  Interventions: Drug: Ocular lubricant

INTERVENTIONS:
Device: Intense pulsed light — Intense pulsed light exerts photothermal, photochemical effects, and photobiomodulation on meibomian glands.
  Arms: IPL arm
Device: thermal pulsation therapy — Thermal pulsation therapy utilizes local heating and massage on the eyelids.
  Arms: TPT arm
Drug: Ocular lubricant — Ocular lubricants moisturize the ocular surface.
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to understand novel treatment methods for meibomian gland dysfunction (MGD)-associated dry eye disease (DED) by comparing two treatment modalities- intense pulsed light (IPL) and thermal pulsation therapy (TPT), to find out the difference of their therapeutic mechanisms and treatment effects, so that eye doctors can give more precise advice to the patients when making treatment decisions.

The main questions it aims to answer are:

* What subtype of meibomian gland dysfunction (MGD) better responds to which treatment modality?
* How long do the treatment effects last?

Researchers will compare each group (IPL and TPT) to a control group treated with eyedrops.

* Do combined treatment of IPL or TPT with eyedrops show better outcomes than only eyedrops?

Participants will:

* Receive different treatment for 2 months according to the group they were randomly allocated to.
* Visit the clinic for checkups after 1 and 3 months after completing the treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with meibomian gland dysfunction (MDG)-associated dry eye disease (DED) that are suitable for intense pulsed light (IPL) and thermal pulsation therapy (TPT)

Exclusion Criteria:

* ocular surgery or trauma in the recent 3 months
* ocular infection
* eyelid abnormalities (e.g., entropion, ectropion, lagophthalmos, severe ptosis or trichiasis)
* blepharospasm
* eyelid tumor
* severe meibomian gland atrophy
* allergic to topical anesthetics
* sunbathe in recent one month
* periocular fillers

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) questionnaire | From enrollment to the end of post-treatment follow-up at 5 months.
  Ocular Surface Disease Index (OSDI) questionnaire was assessed by participants in each follow-ups.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biophotonics, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided